CLINICAL TRIAL: NCT05241678
Title: Study Title: Evaluation of the 24/7 EEG™ SubQ System in Subjects With Uncontrolled Genetic Generalised Epilepsy Syndrome
Brief Title: Evaluation of the 24/7 EEG™ SubQ System in Subjects With Uncontrolled Genetic Generalised Epilepsy Syndrome
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: UNEEG Medical A/S (Industry); Science Foundation Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 20-011
Record Dates: First submitted 2021-11-22; First posted 2022-02-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy, Generalized
MeSH Terms: conditions — Epilepsy, Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a 12 week prospective, comparative investigation in subjects diagnosed with uncontrolled genetic generalised epilepsy (GGE) also known as idiopathic generalised epilepsy (IGE). The purpose of the study is to evaluate whether the 24/7 EEG™ SubQ system, a subcutaneous implantable device, will demonstrate seizure sensitivity approximating that of inpatient video-EEG monitoring with the standard 10-20 electrode system.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of the '24/7 EEG SubQ system' monitoring device in uncontrolled generalised genetic epilepsy syndromes. It is hypothesised that this system will demonstrate seizure sensitivity comparable to Video EEG monitoring with a standard 10-20 electrode system, which is done in a hospital setting and is considered the gold standard for a diagnosis/evaluation of epilepsy.

Ten patients will be recruited with uncontrolled genetic generalised epilepsy. All adults between ages 18-75 years with the ability to give full informed consent. This is an subcutaneously implanted ambulatory device; we will record EEG over a period of twelve weeks. The device consists of two parts: an implant - UNEEG - and an external storage unit (ELG) x 2 that also powers up the implant wirelessly through an inductive link. When the two parts are aligned on opposite sides of the skin: an external pad sits over the implanted device and EEG is recorded from the implanted contacts.

The device is inserted under local anaesthetic by a neurosurgeon subcutaneously overlying the temporal region.

Seizures will be recorded for 12 weeks, then the device will be removed. During the recording period, the patient will undertake video EEG monitoring with the aim of diagnosing seizures by video EEG (gold standard for diagnosis) and comparing the video EEG data with the UNEEG-recorded data.

Throughout the recording period the patients will be overseen by their neurology team.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of refractory genetic generalised epilepsy. Refractory: failure of 2 or more AEDs at appropriate dose.

Seizure frequency of at least one per month over the past 18 months. Subject willing and able to give written informed consent. Subject or guardian has ability to operate system. Subject is able and willing to complete all investigations, required procedures, assessments and follow up.

Subject will tolerate a planned EMU admission within 4 weeks of insertion of device.

Exclusion Criteria:

Subjects who lack capacity to give fully informed consent. Candidates must be at no risk of surgical complications - on no more than 2 days per week of chemotherapy, blood thinning agents, or NSAID.

Device is non-MRI compatible; subjects should not be scheduled for MRI after enrolment, operate or be near an MRI scanner.

Contraindication to use of local anaesthetic drugs during implant and explant surgery.

Pregnancy. Activities that might infer additional risk at participation or affect quality of data. Subject has a hobby or job that delivers extreme pressure variations, ie, diving (5metres acceptable), or that imposes risk or trauma for the device, ie boxing.

Skeletal deformity at insertion site, impeding correct electrode placement. Existing infection at insertion site Participant has or is exposed to a medical device that delivers electrical current near the area of implant - DBS, cochlear implant. VNS is not excluded.

Previous surgery not an exclusion criteria Subjects scheduled for the following treatments within 4 weeks of enrolment: MRI, radiotherapy, U/S close to implant site, ECT, electro knife procedures.

Subject unable or does not have the assistance to operate the device properly.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Beaumont Hospital neurology patients with refractory generalised genetic epilepsy. Consenting adults between the ages of 18/75 yrs, with full capacity
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Electrographic seizure recording sensitivity of the 24/7 EEG™ SubQ system: proportion of identified seizures as compared to ipsilateral video-EEG recordings with the standard 10-20 electrode system. | 12 weeks
  Electroclinical seizure count recorded on SubQ EEG compared to vEEG.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Delanty, MD, Principal Investigator — Royal College of Surgeons, Dublin, Ireland
Locations (1):
- RCSI, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No